CLINICAL TRIAL: NCT05207527
Title: Design and Effectiveness of Different Physical Exercise-based Interventions About Health Indicators and Quality of Life in Patients With Chronic Kidney Disease in Hemodialysis
Brief Title: Intradialisis Physical Exercise in Quality of Life and Health
Acronym: EJERINTRA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Rosario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DVO005 769-CV1091
Record Dates: First submitted 2021-09-22; First posted 2022-01-26 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic kidney disease; Health indicators; Quality of life; Hemodialysis; Peritoneal dialysis; Cardiovascular exercise; Resistance exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Muscle Strength

STUDY DESIGN:
Intervention Model Description: There will be 4 parallel groups, 3 intervention and 1 control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants will be randomized; however, since it is an exercise intervention, the participants cannot be masked. When the interpretation of the data is performed, the researcher will not know what type of treatment the person being evaluated is receiving, and the researcher's advisor will make the comparison without knowing what intervention the participant was subjected to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cardiovascular exercise (Experimental): Cycloergometer
  Interventions: Other: cardiovascular exercise
- Muscle strength (Experimental): Strength exercises will be performed during the hemodialysis session.
  Interventions: Other: Muscle strength
- Mixed (Experimental): Both aerobic and muscular strength exercises will be performed.
  Interventions: Other: cardiovascular exercise; Other: Muscle strength; Other: Mixed
- Control (No Intervention): Conventional treatment or dyalisis usual care

INTERVENTIONS:
Other: cardiovascular exercise — Exercise that mainly stimulates the cardiovascular and respiratory systems.
  Other Names: No aplicable
  Arms: Cardiovascular exercise; Mixed
Other: Muscle strength — Exercise that primarily stimulates the musculoskeletal system.
  Other Names: No aplicable
  Arms: Mixed; Muscle strength
Other: Mixed — Exercise that stimulates the musculoskeletal, cardiovascular and respiratory systems.
  Other Names: No aplicable
  Arms: Mixed

SUMMARY:
Evaluate the effectiveness of different modalities of physical exercise about clinical health indicators and quality of life of patients with chronic kidney disease undergoing hemodialysis.

DETAILED DESCRIPTION:
Objective of this study will be evaluate the effectiveness of different modalities of physical exercise about clinical health indicators and quality of life of patients with chronic kidney disease undergoing on hemodialysis. This study will include to 100 people over 18 years old who are stage five of chronic kidney disease and go to hemodialysis units of Bogota D.C, Colombia.

The ransomized controlled clinical trial to clusters, with 3 groups of intervetion and 1 control, double masking. All the participants receive information on informed consent. The study was approved by the ethics committee of the Universidad del Rosario

ELIGIBILITY:
Inclusion Criteria:

* Include participants with stage five of chronic kidney disease,
* People over 18 years old.
* Their participation is voluntary and their have signed the informed consent form.
* Persons that are undergoing hemodialysis for at least 3 months.
* Persons have ability to do exercise protocols.
* Persons have the approval by nephrologist doctor and deportologist for to do the study according to the results of initial medical assessment.

Exclusion Criteria:

* Surgical intervention to least 6 months.
* Skeletal limitations that affect exercise performance.
* Psychiatric disorders and psychological such as depression, anxiety that could be affect participation of the study.
* Body Mass Index greater than 30 kg/m2 and not less than 18.5 kg/m2.
* Hemodialysis catheter dysfunction or infection as well as participation in home exercise programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2028-10-12 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Health indicators - Dialysis efficiency | 6 months
  Dialysis efficiency will be measured by analysis through biochemical methods in blood serum (KT/V).
Health indicators - KT/V | 6 months
  It is an indicator of the rate of clearance of urea and other wastes by the dialyzer.
Health indicators - Sarcopenia | 6 months
  Sarcopenia will be measured by means of dynamometry, in the upper limb it will be evaluated using a handgrip dynamometer Participants will be instructed to stand with their arms fully extended by gradually and continuously squeezing their grip until they reach their maximum strength for at least 2 seconds, the test will be performed twice. In lower limb will be performed by means of lower limb dynamometer in which the subject holds the center of the bar, palms down, head straight and back straight, flexes the knees at an angle of 120° and the length of the chain is adjusted so that the bar is in the crease formed between the thigh and the trunk. The subject can place his hands in the middl
Kidney Disease and Quality of Life (KDQOL-36) | 6 months
  This will be measured by means of the Kidney Disease and Quality of Life Questionnaire (KDQOL-36) which is defined as a specific questionnaire for patients with kidney disease on dialysis, developed by the Kidney Disease Quality of Life Working Group as a specific self-report measure of health-related quality of life or perceived health in these individuals. It is a self-report questionnaire that combines the generic SF-36 health survey instrument and disease-specific components to assess the health-related quality of life of patients with chronic kidney disease. The minimum value is 0 and the maximum value is 100. A higher score means a better quality of life
Physical condition - Body composition1 | 6 months
  This variable will be measured by means of bioimpedance, which is defined as a non-invasive method, where the electrical properties of the human body are used to estimate body water and the different body tissues, obtaining results in percentage of body mass index, visceral fat percentage, total body fat and muscle percentage.
Physical condition - Body composition2 | 6 months
  This variable will be measured by means of bioimpedance, which is defined as a non-invasive method, where the electrical properties of the human body are used to estimate body water and the different body tissues, obtaining results in percentage of body mass index.
Physical condition - Body composition3 | 6 months
  This variable will be measured by means of bioimpedance, which is defined as a non-invasive method, where the electrical properties of the human body are used to estimate body water and the different body tissues, obtaining results in percentage of visceral fat percentage.
Physical condition - Body composition4 | 6 months
  This variable will be measured by means of bioimpedance, which is defined as a non-invasive method, where the electrical properties of the human body are used to estimate body water and the different body tissues, obtaining results in percentage of total body fat.
Physical condition - Body composition5 | 6 months
  This variable will be measured by means of bioimpedance, which is defined as a non-invasive method, where the electrical properties of the human body are used to estimate body water and the different body tissues, obtaining results in body muscle percentage.
Muscle strength | 6 months
  The muscle strength will be measured by means of dynamometry, in the upper limb it will be evaluated using a handgrip dynamometer Participants will be instructed to stand with their arms fully extended by gradually and continuously squeezing their grip until they reach their maximum strength for at least 2 seconds, the test will be performed twice. In lower limb will be performed by means of lower limb dynamometer in which the subject holds the center of the bar, palms down, head straight and back straight, flexes the knees at an angle of 120° and the length of the chain is adjusted so that the bar is in the crease formed between the thigh and the trunk. The subject can place his hands in the middl
Fatigue | 6 months
  This variable will be measured by means of the Fatigue Severity Scale created by Krupp for the assessment of fatigue. It consists of 9 items with a Likert-type response with 7 possibilities, of increasing intensity and scoring between 1 and 7, the total is given with the sum of all items. Its objective is to determine the severity of fatigue in patients with renal disease.
Functional capacity - SPPB | 6 months
  This variable will be measured by means of a questionnaire called Short Physical Performance Battery. The purpose of this test is to evaluate the functioning of the lower extremities in the elderly and it is applied to older adults who have the ability to transfer from sitting to standing autonomously and without the help of the upper limbs.
Functional capacity -6MWT | 6 months
  The functional capacity will also be measured by means of the 6-minute test, which is defined as a constant load stress test that measures the distance a person can walk in a period of six minutes, at a fast pace, on a flat, hard surface.
Functional capacity - 2MT | 6 months
  The functional capacity will also be measured by means of the two-minute stationary gait test, which consists of the individuals evaluated marching in place as fast as possible for 2 minutes; reference values have been published for adults between 60 and 94 years of age.

SECONDARY OUTCOMES:
Depression and anxiety (Beck Scale) | 6 months
  This will be measured by means of the Beck Depression and Anxiety Scale. It is a self-assessment scale that primarily assesses the clinical symptoms of melancholy and intrusive thoughts present in depression.
  It is the one with the highest percentage of cognitive symptoms, highlighting also the absence of motor and anxiety symptoms. It is commonly used to assess the severity of the disease. Scale values range from 0 to 63, a higher score represents a worse outcome.

OTHER OUTCOMES:
Caloric intake | 6 months
  Measured by means of the intake diary
Number of participants that Smoke | 6 months
  Assessed by means of surveys. Absence or presence of smoking habit
Prevalence of hemodialysis | 6 months
  Assessed by clinical history.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Ramos-Caballero, CI, Study Chair — Universidad del Rosario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan D, Cheema BS. Progressive Resistance Training in End-Stage Renal Disease: Systematic Review. Am J Nephrol. 2016;44(1):32-45. doi: 10.1159/000446847. Epub 2016 Jun 30. PMID 27355619
- [Background] Chung YC, Yeh ML, Liu YM. Effects of intradialytic exercise on the physical function, depression and quality of life for haemodialysis patients: a systematic review and meta-analysis of randomised controlled trials. J Clin Nurs. 2017 Jul;26(13-14):1801-1813. doi: 10.1111/jocn.13514. Epub 2017 Mar 20. PMID 27532211
- [Background] Ferrari F, Helal L, Dipp T, Soares D, Soldatelli A, Mills AL, Paz C, Tenorio MCC, Motta MT, Barcellos FC, Stein R. Intradialytic training in patients with end-stage renal disease: a systematic review and meta-analysis of randomized clinical trials assessing the effects of five different training interventions. J Nephrol. 2020 Apr;33(2):251-266. doi: 10.1007/s40620-019-00687-y. Epub 2019 Dec 21. PMID 31865607
- [Background] Molsted S, Bjorkman ASD, Lundstrom LH. Effects of strength training to patients undergoing dialysis: a systematic review. Dan Med J. 2019 Jan;66(1):A5526. PMID 30573007
- [Background] Pu J, Jiang Z, Wu W, Li L, Zhang L, Li Y, Liu Q, Ou S. Efficacy and safety of intradialytic exercise in haemodialysis patients: a systematic review and meta-analysis. BMJ Open. 2019 Jan 21;9(1):e020633. doi: 10.1136/bmjopen-2017-020633. PMID 30670499
- [Background] Scapini KB, Bohlke M, Moraes OA, Rodrigues CG, Inacio JF, Sbruzzi G, Leguisamo CP, Sanches IC, Tourinho Filho H, Irigoyen MC. Combined training is the most effective training modality to improve aerobic capacity and blood pressure control in people requiring haemodialysis for end-stage renal disease: systematic review and network meta-analysis. J Physiother. 2019 Jan;65(1):4-15. doi: 10.1016/j.jphys.2018.11.008. Epub 2018 Dec 21. PMID 30581137
- [Background] Young HML, March DS, Graham-Brown MPM, Jones AW, Curtis F, Grantham CS, Churchward DR, Highton P, Smith AC, Singh SJ, Bridle C, Burton JO. Effects of intradialytic cycling exercise on exercise capacity, quality of life, physical function and cardiovascular measures in adult haemodialysis patients: a systematic review and meta-analysis. Nephrol Dial Transplant. 2018 Aug 1;33(8):1436-1445. doi: 10.1093/ndt/gfy045. PMID 29608708
- [Background] Afsar B, Siriopol D, Aslan G, Eren OC, Dagel T, Kilic U, Kanbay A, Burlacu A, Covic A, Kanbay M. The impact of exercise on physical function, cardiovascular outcomes and quality of life in chronic kidney disease patients: a systematic review. Int Urol Nephrol. 2018 May;50(5):885-904. doi: 10.1007/s11255-018-1790-4. Epub 2018 Jan 17. PMID 29344881
- [Background] Andrade FP, Rezende PS, Ferreira TS, Borba GC, Muller AM, Rovedder PME. Effects of intradialytic exercise on cardiopulmonary capacity in chronic kidney disease: systematic review and meta-analysis of randomized clinical trials. Sci Rep. 2019 Dec 5;9(1):18470. doi: 10.1038/s41598-019-54953-x. PMID 31804617
- [Background] Bohm J, Monteiro MB, Andrade FP, Veronese FV, Thome FS. Acute effects of intradialytic aerobic exercise on solute removal, blood gases and oxidative stress in patients with chronic kidney disease. J Bras Nefrol. 2017 Apr-Jun;39(2):172-180. doi: 10.5935/0101-2800.20170022. Epub 2017 Apr 27. English, Portuguese. PMID 28489182
- [Background] Anding K, Bar T, Trojniak-Hennig J, Kuchinke S, Krause R, Rost JM, Halle M. A structured exercise programme during haemodialysis for patients with chronic kidney disease: clinical benefit and long-term adherence. BMJ Open. 2015 Aug 27;5(8):e008709. doi: 10.1136/bmjopen-2015-008709. PMID 26316654
- [Background] Clarkson MJ, Bennett PN, Fraser SF, Warmington SA. Exercise interventions for improving objective physical function in patients with end-stage kidney disease on dialysis: a systematic review and meta-analysis. Am J Physiol Renal Physiol. 2019 May 1;316(5):F856-F872. doi: 10.1152/ajprenal.00317.2018. Epub 2019 Feb 13. PMID 30759022
- [Background] Salhab N, Karavetian M, Kooman J, Fiaccadori E, El Khoury CF. Effects of intradialytic aerobic exercise on hemodialysis patients: a systematic review and meta-analysis. J Nephrol. 2019 Aug;32(4):549-566. doi: 10.1007/s40620-018-00565-z. Epub 2019 Jan 18. PMID 30659520
- [Background] Smart N, Steele M. Exercise training in haemodialysis patients: a systematic review and meta-analysis. Nephrology (Carlton). 2011 Sep;16(7):626-32. doi: 10.1111/j.1440-1797.2011.01471.x. PMID 21557787
- [Background] Tentori F, Elder SJ, Thumma J, Pisoni RL, Bommer J, Fissell RB, Fukuhara S, Jadoul M, Keen ML, Saran R, Ramirez SP, Robinson BM. Physical exercise among participants in the Dialysis Outcomes and Practice Patterns Study (DOPPS): correlates and associated outcomes. Nephrol Dial Transplant. 2010 Sep;25(9):3050-62. doi: 10.1093/ndt/gfq138. Epub 2010 Apr 13. PMID 20392706
- [Background] Silva SF, Pereira AA, Silva WA, Simoes R, Barros Neto Jde R. Physical therapy during hemodialyse in patients with chronic kidney disease. J Bras Nefrol. 2013 Jul-Sep;35(3):170-6. doi: 10.5935/0101-2800.20130028. English, Portuguese. PMID 24100735
- See also: Fisioterapia durante la hemodiálisis: resultados de un programa de fuerza-resistencia — http://revistanefrologia.com/es-fisioterapia-durante-hemodialisis-resultados-un-programa-fuerza-resistencia-articulo-X0211699508033146
- See also: Beneficios del ejercicio físico de baja intensidad durante la sesión de hemodiálisis en el paciente anciano — http://www.revistanefrologia.com/es-beneficios-del-ejercicio-fisico-baja-articulo-S0211699515000685
- See also: Factores no tradicionales influyentes en la calidad de vida de los pacientes de hemodiálisis — http://revistanefrologia.org/index.php/rcn/article/view/147?source=/index.php/rcn/article/view/147